CLINICAL TRIAL: NCT00355108
Title: ATERO : A Randomised Study With Tranexamic Acid in Epistaxis of Rendu Osler Syndrome. Beneficial or Iatrogenic Effects.
Brief Title: ATERO : A Randomised Study With Tranexamic Acid in Epistaxis of Rendu Osler Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Henri PLAUCHU, MD, Hospices Civils de Lyon
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2005.405
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2010-12

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic; Osler-Rendu Disease
Keywords: Rendu Osler syndrome; Epistaxis; Tranexamic acid; clinical trial
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tranexamic acid — 2 3-month-periods in cross-over: placebo or 3g/day of tranexamic acid

SUMMARY:
Scientific Objectives Primary objective : Demonstrate that oral intake of tranexamic acid significantly reduces the risk of epistaxis occurrence, estimated by the average monthly duration of episodes of epistaxis.

Secondary objectives :

* Document the benefit of tranexamic acid on the amount of haemoglobine and quality of life of patients.
* Identify scalable and genetic factors of response to the treatment by tranexamic acid.
* Describe compliance and tolerance of the treatment. Method Experimental Design We suggest the realisation of a randomised comparative clinical trial versus placebo, with a crossover of random alternated periods of three months over a total of six months.

Study Population 213 affected patients, displaying sufficiently invalidating epistaxis to require a basal treatment, will be recruited and followed every 3 months. Recruitment will lean on teams who are part of the national French network in close collaboration with the reference centre for the Rendu-Osler disorder, appointed to Lyon on the 19th of November 2004. Follow up of the study will be carried out by the Clinical Investigational Centre of the related towns.

Outcome measures The main criterion of efficacy is the average duration of epistaxis, the secondary criterion of efficacy is the average number of epistaxis measured per month. Tolerance will be analysed according to the occurrence of venal or arterial thrombosis and allergic accidents. Venal thrombosis will systematically be sought by an inferior limbs echodoppler. Response markers will be sought through modelisation incorporating environmental, phenotypic and genetic factors.

DETAILED DESCRIPTION:
Argumentation Rendu-Osler syndrome, rare but ubiquitary, affects at least 8000 persons in France. This genetic disorder is characterised by a dominant autosomal hereditary transmission of telangiectasis and arteriovenous fistulae. The most apparent expression of the disorder, often the cause of chronic anaemia, is the occurrence of spontaneous, repeated, frequent and sometimes abundant epistaxis to the extent that continuous martial treatment and multiple transfusions are necessary. The handling of this major symptom of the disorder is badly coded and often demands local ENT treatments or medication whose efficacy is not sufficiently documented. Among them, an anti-fibrinolytic, tranexamic acid, has been evaluated several times with a low level of proof, so that it is regularly prescribed with a good impression of efficacy for certain patients. It therefore seems essential that these prescriptions should be based on more reliable data thereby providing clearer information to patients regarding the expected benefits. The recent report of a high frequency of thrombophlebitis in RO patients and the ancient concept of coagulation disorders or thrombosis (Bick 1981) have lead to a restriction of the inclusion criteria and a systematic search for a possible iatrogenic effect (inferior limbs venous echodoppler).

Scientific Objectives Primary objective : Demonstrate that oral intake of tranexamic acid significantly reduces the risk of epistaxis occurrence, estimated by the average monthly duration of episodes of epistaxis.

Secondary objectives :

* Document the benefit of tranexamic acid on the amount of haemoglobine and quality of life of patients.
* Identify scalable and genetic factors of response to the treatment by tranexamic acid.
* Describe compliance and tolerance of the treatment. Method Experimental Design We suggest the realisation of a randomised comparative clinical trial versus placebo, with a crossover of random alternated periods of three months over a total of six months.

Study Population 213 affected patients, displaying sufficiently invalidating epistaxis to require a basal treatment, will be recruited and followed every 3 months. Recruitment will lean on teams who are part of the national French network in close collaboration with the reference centre for the Rendu-Osler disorder, appointed to Lyon on the 19th of November 2004. Follow up of the study will be carried out by the Clinical Investigational Centre of the related towns.

Outcome measures The main criterion of efficacy is the average duration of epistaxis, the secondary criterion of efficacy is the average number of epistaxis measured per month. Tolerance will be analysed according to the occurrence of venal or arterial thrombosis and allergic accidents. Venal thrombosis will systematically be sought by an inferior limbs echodoppler. Response markers will be sought through modelisation incorporating environmental, phenotypic and genetic factors.

Expected benefits From an individual point of view, the knowledge of the response to tranexamic acid measured the most precisely possible, represents a benefit for each study participant, who will be able to continue the treatment knowingly if it proves efficient. From a general point of view, the ATERO study will aid in the decision whether to continue this course of action which despite its lack of proof is justified by its efficacy as well as its cost and absence of adverse effects. The precise documentation of its innocuousness may be necessary by the means of a specific study depending on the results on the ATERO study.

ELIGIBILITY:
Inclusion Criteria:

* Repeated, spontaneous epistaxis in a known Rendu Osler patient who wants global caring, these must be daily epistaxis (> 28 a month) or a total amount of 60 minutes of bleeding a month (50 % Rendu-Osler patients bleed before 20 and 99 % at 50 when penetrance is complete).
* Good completion of the grid of control by recording the number and duration of epistaxis over a period of three month.

Exclusion Criteria:

* Rendu Osler syndrome with specific phenotype : absence of epistaxis or occasional epistaxis, no need for particular care.
* Maintained expectations of an ENT treatment of epistaxis in a delay of three months.
* Incapacity of detailing the number of epistaxis, especially, at least, within three months before entering the study.
* No informed consent obtained after informing the patient on his participation to the study.
* Expected lack of observance because of an incapacity to compel to the daily treatment.
* Formal indication to Tranexamic Acid (angioneurotic oedema as a disease modifying treatment of 3 to 4 g/ day).
* Contra-indications to Tranexamic acid: history of convulsion, arterial or veinous thrombosis, , positivity of veinous echo doppler of the inferior limbs; Serum creatinine > 250 µmol/l.

N.B. Cases of bad observance are not frequent, patients being highly concerned with a treatment to reduce their discomfort and anaemia. They are more likely ready to move to a centre insuring this handling. Nevertheless, lack of observance will be detected over a period of 15 days of placebo in simple blind, before randomization.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2006-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy criterion is the average monthly duration of epistaxis. | after first 3 month period treatment or placebo and after second 3 month period treatment or placebo

SECONDARY OUTCOMES:
the average monthly number of epistaxis, | after first 3 month period treatment or placebo and after second 3 month period treatment or placebo
the average duration of one episode of epistaxis measured over a month, | after first 3 month period treatment or placebo and after second 3 month period treatment or placebo
the Haemoglobin level | after first 3 month period treatment or placebo and after second 3 month period treatment or placebo
estimation of Quality of life. | over first 3 month period treatment or placebo and over second 3 month period treatment or placebo
Outcome of following Adverse Event: arterial or veinous thrombosis, allergic accident | during first 3 month period treatment or placebo and over second 3 month period treatment or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Henri PLAUCHU, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Henri PLAUCHU, Lyon, France

REFERENCES:
- [Result] Gaillard S, Dupuis-Girod S, Boutitie F, Riviere S, Moriniere S, Hatron PY, Manfredi G, Kaminsky P, Capitaine AL, Roy P, Gueyffier F, Plauchu H; ATERO Study Group. Tranexamic acid for epistaxis in hereditary hemorrhagic telangiectasia patients: a European cross-over controlled trial in a rare disease. J Thromb Haemost. 2014 Sep;12(9):1494-502. doi: 10.1111/jth.12654. Epub 2014 Jul 29. PMID 25040799